CLINICAL TRIAL: NCT00414895
Title: Absolute Myocardial Perfusion Measurement in the Transplanted Heart: a New Method for Accurate Detection of Allograft Rejection. A Pilot Study
Brief Title: Absolute Myocardial Perfusion Measurement in the Transplanted Heart
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other); Swiss Heart Foundation (Other)
Responsible Party: Christian Seiler, MD, Professor and Co-Chairman of Cardiology, Department of Cardiology, University Hospital, CH-3010 Bern, Switzerland
Other Study IDs: 216/06
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Cardiac Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The goal of this study is to detect AR and CR in the transplanted heart by quantitative assessment of myocardial blood flow and its constituents by myocardial contrast echocardiography (MCE). Further we investigate the collateral circulation in these patients.

DETAILED DESCRIPTION:
Heart transplantation has become an accepted therapy for end-stage heart failure. Acute allograft rejection (AR) remains a major cause of mortality in heart transplant recipients. Chronic rejection (CR) determines the long-term prognosis after cardiac transplantation and is responsible for more than one third of late deaths. Different non-invasive methods have been evaluated for the detection of AR, but the gold standard remains endomyocardial biopsy (EMB).

Very little is known about the impact of CR on the collateral circulation in transplant patients. Since the collateral circulation of the heart is mainly part of the microcirculation, it can be hypothesized that it is less developed than in "normal" coronary atherosclerosis without microvascular lesions.

The quantification of CR with non-invasive techniques has remained difficult. In this context, there is a need for a reliable non-invasive test to avoid regularly invasive evaluation.

Based on the above considerations we propose that both AR and CR can be accurately detected and differentiated using non-invasive quantitative myocardial contrast echocardiography (MCE).

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart transplantation, age 18-82 years
* EMB or EMB and coronary angiography
* Written informed consent to participate in the study

Exclusion Criteria:

* Known adverse reaction to adenosine or echo contrast (SonoVueâ)
* Second or third degree AV block, unprotected sick sinus syndrome, atrial fibrillation with uncontrolled ventricular rate
* Asthma, severe pulmonary arterial hypertension (systolic pulmonary artery pressure >50mmHg assessed by echocardiography)
* Severe obstructive pulmonary disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective study with consecutive inclusion of transplanted patients undergoing follow-up exams. Examinations comprise endomyocardial biopsy (EMB) and, partly, coronary angiography on the subsequent day. Group A patients (i.e. those without coronary angiography) undergo MCE and pharmacologic stress with adenosine, the results of which are compared with the EMB done at the same day. If they have an acute rejection, they are reexamined during a histologically proven rejection free period, and the results are compared with those obtained during acute rejection. Group B patients (i.e. with EMB and coronary angiography) undergo the same procedure as in group A. Additionally, coronary collateral flow index (CFI) is obtained and an IVUS exam is performed during coronary angiography.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, Prof., Principal Investigator — University Hospital Bern, Switzerland
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

REFERENCES:
- [Derived] Rutz T, de Marchi SF, Roelli P, Gloekler S, Traupe T, Steck H, Eshtehardi P, Cook S, Vogel R, Mohacsi P, Seiler C. Quantitative myocardial contrast echocardiography: a new method for the non-invasive detection of chronic heart transplant rejection. Eur Heart J Cardiovasc Imaging. 2013 Dec;14(12):1187-94. doi: 10.1093/ehjci/jet066. Epub 2013 Apr 23. PMID 23612502